CLINICAL TRIAL: NCT06094452
Title: Effects of 24-week Computerized Cognitive Training on Microbiota-gut-brain Axis in Patients With Mild Cognitive Impairment and Mild Alzheimer's Disease: a Randomized Controlled Trial
Brief Title: Effects of 24-week Computerized Cognitive Training in Patients With MCI and AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Wenbo Zhang, Principle Investigator, Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChongqingMU9
Record Dates: First submitted 2023-10-04; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
Keywords: computerized cognitive training; functional near-infrared spectroscopy; mild cognitive impairment; Alzheimer's disease; brain-gut-microbiota axis; gut microbiota
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: After recruitment and baseline assessments, pairs of participants with MCI and mild AD will be randomly allocated into either the CCT group and the control group. Participants in CCT group will receive a multidomain adaptive computerized cognitive training program (www.66nao.com) for 24 weeks. Patients in control group will receive treatment as usual (TAU) for 24 weeks.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Since it will not be possible to blind the participants because the experimental and control interventions have to be explained to them and their caregivers before randomization. The single blinding will be applied to researchers who conducted the measurements to minimize the potential assessor biases. Blinding will be also maintained for data management, outcome assessment, and data analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerized Cognitive Training (Experimental): Adaptive computerized cognitive training program (www.66nao.com) and the intensity is at least 30 minutes of training per day (3 cycle of 5 2-min tasks), 5 days a week for 24 weeks.
  Interventions: Other: Computerized Cognitive Training
- Treatment As Usual (Active Comparator): Patients in control group will receive TAU for 24 weeks, which includes (1) regular medication management from the Memory Clinic, if applicable; (2) basic health education at each follow-up (face to face) and twice per month on the internet.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Other: Computerized Cognitive Training — Participants in intervention group will receive a multidomain, adaptive computerized cognitive training program (www.66nao.com) and will be required to complete at least 30 minutes of training per day (3 cycle of 5 2-min tasks), 5 days a week for 24 weeks. Multidomain coverage paradigms include working memory, calculation, processing speed, attention, executive function, and short-term and long-term memory.
  Arms: Computerized Cognitive Training
Other: Treatment As Usual — Patients in control group will receive TAU for 24 weeks, which includes (1) regular medication management from the Memory Clinic, if applicable; (2) basic health education at each follow-up (face to face) and twice per month on the internet .
  Arms: Treatment As Usual

SUMMARY:
This study aims to testify multi-domain effects of computerized cognitive training in patients with mild cognitive impairment and mild Alzheimer's disease through multi-dimensional evaluation.

DETAILED DESCRIPTION:
This study aimed to elucidate the neural process enhancement and remodulation in gut microbes resulting from older adults with MCI and mild AD in a randomized controlled trial of a 24-week computerized cognitive training (CCT) program.

After recruitment and baseline assessments, pairs of participants with MCI and mild AD would be randomly allocated into the corresponding subgroup. Participants in CCT group will receive a computerized multidomain cognitive training program (www.66nao.com) and will be required to complete at least 30 minutes of training per day (3 cycle of 5 2-min tasks), 5 days a week for 24 weeks. Adherence to the intervention will be supervised by an independent researcher. The number of training days and training hours per day will be recorded. Patients in control group received treatment as usual (TAU) for 24 weeks. The neuropsychological measures will be performed at baseline, follow-up at 4 weeks, 12 weeks, and 24 weeks; functional Near-Infrared Spectroscopy (fNIRS) data and fecal samples will collected at baseline and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* between 55 and 90 years of age;
* a Clinical Dementia Rating (CDR) score of 0.5 or 1;
* at least three months of stable doses if receiving antidementia medication or mood-stabilizing medication for mild AD participants;
* primary school education and above;
* accompanied by a consistent caregiver (at least 5 days/week);
* informed consent.

Exclusion Criteria:

* factors that might preclude completion of assessments;
* severe psychiatric illness and the use of antidepressants;
* any condition that would preclude completion of training and follow-up tests;
* other disorders that would affect cognition.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Global Cognition | baseline, 4, 12, 24 weeks
  The Alzheimer's Disease Assessment Scale- cognitive subscale (11 items) will be used to evaluate global cognition and served as the primary outcome measure. The minimum and maximum values are 0 and 70 respectively, and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Learning | baseline, 4, 12, 24 weeks
  The Auditory Verbal Learning Test (minimum to maximum: 0-45) will be applied, and higher scores mean a better outcome for the scale.
Episodic Memory | baseline, 4, 12, 24 weeks
  The Free and Cued Selective Reminding Test (minimum to maximum: 0-48) will be applied, and higher scores mean a better outcome for the scale.
Attention | baseline, 4, 12, 24 weeks
  The Trail Making Test (minimum to maximum: 0-24) will be applied, and higher scores mean a better outcome for the scale.
Executive Function | baseline, 4, 12, 24 weeks
  The Digital Span Test (minimum to maximum: 0-10) will also be applied, and higher scores mean a better outcome for the scale.
Visuospatial Function | baseline, 4, 12, 24 weeks
  The Clock Drawing Test (minimum to maximum: 0-15) will be applied, and higher scores mean a better outcome for the scale.
Verbal Ability | baseline, 4, 12, 24 weeks
  The Boston Naming Test (minimum to maximum: 0-30) will be applied, and higher scores mean a better outcome for the scale.
Verbal Frequency | baseline, 4, 12, 24 weeks
  The Verbal Frequency Test (minimum: 0, no maximum) will also be applied, and higher scores mean a better outcome for the scale.
Neuropsychiatric Symptoms | baseline, 4, 12, 24 weeks
  The Neuropsychiatric Inventory (minimum to maximum: 0-144) will be used, and higher scores mean a worse outcome for the scale.
Depression | baseline, 4, 12, 24 weeks
  The 30-Geriatric Depression Scale (minimum to maximum: 0-30) will be used, and higher scores mean a worse outcome for the scale.
Daily Living Function | baseline, 4, 12, 24 weeks
  The Instrumental Activities of Daily Living scale (minimum to maximum: 0-31) will be used, and higher scores mean a worse outcome for this scale.
Severity of Cognitive Impairment | baseline, 4, 12, 24 weeks
  The Clinical Dementia Rating scale (sum of boxes, minimum to maximum: 0-18) will be used, and higher scores mean a worse outcome for this scale.
Brain Functional Connectivity | baseline and 24 weeks
  The regions of interests (ROIs) are selected as the Brodmann Area (BA) 9 and 46 (overlapping the dorsolateral prefrontal cortex, DLPFC), left Brodmann Area 6 (overlapping pre-Motor and Supplementary Motor Cortex, PM-SMC), and right Brodmann Area 45 (overlapping pars triangularis Broca's area). For each resting-state dataset of fNIRS, functional connectivity (FC) will be analyzed by Spearman's correlation between the time series of each ROI-to-ROI pair.
Alpha-diversity of Gut Microbiome | baseline and 24 weeks
  Fecal samples will be collected from patients in standard 300 mL sterilin tubes and frozen immediately at -80°C. Patients will be asked to produce the first-morning sample for consistency and to avoid alcohol the previous 24 h. After 16S rRNA high-throughput sequencing, the diversity analysis of species under a sample (α-diversity) of the bacteria on Genus, will be analyzed in R.
Beta-diversity of Gut Microbiome | baseline and 24 weeks
  After 16S rRNA high-throughput sequencing, the cluster analysis between different samples (β-diversity) will be analyzed in R.
Composition of Gut Microbiome | baseline and 24 weeks
  After 16S rRNA high-throughput sequencing, the compositional analysis of bacteria on genus will be analyzed in R.

CONTACTS AND LOCATIONS:
Overall Officials: Weihua Yu, Dr., Principal Investigator — Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
With publication of research articles, de-identified data collected for the study, including individual participant data, can be made available to interested parties on reasonable request, and if in line with privacy regulations. Data can be requested at least 18 months after publication of the research articles, with a proposal by sending an e-mail to Dr. Yang Lü.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data can be requested at least 18 months after publication of the research articles.
Access Criteria: With publication of research articles, de-identified data collected for the study, including individual participant data, can be made available to interested parties on reasonable request, and if in line with privacy regulations, with a proposal by sending an e-mail to Dr. Yang Lü.

REFERENCES:
- See also: The trail has also been registered under chictr.org.cn (ChiCTR2100051362). — http://www.chictr.org.cn/bin/project/edit?pid=125115